CLINICAL TRIAL: NCT00866567
Title: Defects in Opsonophagocytosis in Premature Infants as a Factor for the Development of Neonatal Sepsis
Brief Title: Defects in Opsonophagocytosis in Premature Infants
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Gertrude Von Meissner Foundation (Other); European Society of Intensive Care Medicine (Other); Swiss National Fund for Scientific Research (Other)
Responsible Party: Pierre TISSIERES, MD; MSc, University Hospital, Geneva
Other Study IDs: MatPed 08-017
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2009-03

CONDITIONS: Prematurity; Neonatal Sepsis
Keywords: prematurity; VLBW; sepsis; innate immunity
MeSH Terms: conditions — Premature Birth; Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum cDNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Premature infants of less than 28 weeks of gestational age
- 2: Premature infants of more than 28 weeks and less than 32 weeks of gestational age
- 3: Term newborns
- 4: Adults

SUMMARY:
The purpose of the study is to characterize innate immune function of premature infants, and identify defects that may be responsible for the development of bacterial sepsis.

DETAILED DESCRIPTION:
Sepsis is an important problem in preterm infants and carries a significant morbidity and mortality. It is estimated that 20% of premature infants surviving beyond the first three days of life will have one or more culture-proven bacteremic sepsis. There is increasing epidemiologic and biologic evidence suggesting that preterm newborns are more susceptible to infection than term newborns and adults. Immaturity of the immune system, and, in particular, defects in innate responses to pathogens are of foremost importance in the pathogenesis of neonatal sepsis. The aims of the study are the:

1. Determination of the opsonic capacity of plasma from premature infants, vs. term newborns, and identification possible molecular innate immune defect(s) in preterm plasma.
2. Characterization of the role of TLR2 and TLR4 responses in phagocytes from premature infants using classical TLRs agonists. Determination of the capacity of plasma from premature infants to sustain TLR pathways, with a particular attention paid to the possible role of soluble MD-2 in plasma from premature infants in TLR-dependent opsonophagocytosis.
3. Determine prognostic factors for neonatal sepsis. The identification of a quantitative and/or qualitative defect in innate plasma protein(s) in premature newborns has the potential of identifying those infants who are likely to develop a neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Premature or term delivery

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All premature infants delivered at the University Hospitals of Geneva
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Leukocyte phenotype, opsonophagocytic function, and whole blood response to pathogens | at delivery

SECONDARY OUTCOMES:
Leukocyte phenotype, opsonophagocytic function during neonatal sepsis | 1 week after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Jerome PUGIN, MD, Study Director — University Hospitals of Geneva; Michel BERNER, MD, Study Director — University Hospitals of Geneva; Pierre TISSIERES, MD, MSc, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Geneva 14, Switzerland